CLINICAL TRIAL: NCT00819455
Title: The Role of Information Technology in the Primary Prevention of Type 2 Diabetes
Brief Title: Use of Information Technology in the Prevention of Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: India Diabetes Research Foundation & Dr. A. Ramachandran's Diabetes Hospitals (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Principal Investigator, Dr.A.Ramachandran, President, India Diabetes Research Foundation & Dr. A. Ramachandran's Diabetes Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IT001IDRF-IC
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Prevention of Diabetes; Lifestyle Modification; Text messages
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): In person lifestyle advice at baseline, 6, 12, 18 months.
  Interventions: Behavioral: Control arm (usual care/standard care arm)
- 1 (Experimental): In person lifestyle advice at baseline, 6, 12, 18 months. Receive reminders by internet based, mobile phone text messaging (Frequency, time and number(s) of messages according to participants requirement)
  Interventions: Behavioral: Experimental

INTERVENTIONS:
Behavioral: Experimental — Active Life style modification-motivation by I.T technology
  Arms: 1
Behavioral: Control arm (usual care/standard care arm) — Life style modification only once
  Arms: 2

SUMMARY:
Type 2 diabetes is a major and increasing problem in India and the UK. In clinical trials it can be prevented in people at high risk by lifestyle intervention. While these trials established the proof of principle, they involved a degree of input from healthcare professionals not feasible outside the trial situation. We hypothesize that diabetes prevention can be achieved at lower cost using personalised feedback via mobile phone, based on information on healthy diet and physical activity habits. We shall develop research protocols and computerized algorithms to test this hypothesis in India for application subsequently in the UK and elsewhere.

DETAILED DESCRIPTION:
Diabetes prevention programmes conducted in various ethnic and racial populations have conclusively demonstrated that lifestyle modification (LSM) focussed on caloric restriction and increased physical activity can prevent or postpone the onset of T2DM. The Indian Diabetes Prevention Programme-1 (IDPP-1) conducted by our group established that LSM is an effective tool for the primary prevention of T2DM in Asian Indian subjects (1). But the major hurdle for any clinical trial is to disseminate the intervention principles at a community level is often proved to be very difficult. The main objective of this prevention programme is to determine whether individualized messages on LSM (diet and physical activity) by mobile phone-based message delivery system can help educate and motivate subjects with a high risk for developing type 2 diabetes to adhere to LSM and thereby improve glucose tolerance.

Sample selection:

This is a randomized, controlled prospective study, carried out in participants who have been diagnosed with persistent IGT using the 1999 World Health Organization (WHO) criteria. Interested participants who fulfilled the inclusion criteria participated in this prevention programme. Screening was carried out in the work places. The participants were advised not to do any strenuous work during the screening period. Interested participants, after an overnight fast of 8 to 12 hours, underwent a capillary blood glucose test 2h PG after an ingestion of 75G glucose. Among the subjects identified with IGT, those with 2h PG values >8.9 mmol/l (≥ 160 mg/dl) were invited for a confirmatory OGTT, within a week. During the 2nd GTT, venous blood samples were collected at fasting (0 minute), 30 and 120 minutes after the glucose intake.Subjects who satisfied the criteria for IGT on both occasions were recruited for this prevention programme. Randomized was based on the MATLAB 'randperm' random number generator (MARSAGLIA RANDOM NUMBER generator algorithm).

Recruitment:

Subjects were recruited into two groups:

1. control arm: advised on LSM and the beneficial effects of healthy dietary habits, weight reduction and increased physical activity at the baseline, 6, 12, 18 and 24 months respectively (standard care advise).
2. Intervention group: receive in addition to the above advise would receive frequent text messages on general well being and different forms of physical activity and principles of healthy diet. The frequency and time at which each participant preferred to receive the messages were noted.

Assessments:

Both groups will undergo personal reviews at 6 monthly intervals for a period of 2 years. At randomization, participants were interviewed personally to elicit demographic, medical, diet, behavioral and physical activity details.

6 & 18 month assessments: Diet and physical activity questionnaires, body weight, WC, pulse and BP will be obtained. Two hour post glucose will be measured.

12 & 24 month assessment: Participants will be questioned about the acceptability of the project and its impact on their life. Changes in health will be documented and the physical examination repeated. They will complete further dietary, physical activity and quality of life questionnaires and will be asked about their use of healthcare resources for health economic assessment. The OGTT and ECG will be repeated, with other measurements as at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ≥ 23
* Age ≥ 35 years
* A 1st degree relative with type 2 diabetes

Exclusion Criteria:

* Normal and diabetic subjects
* Presence of other serious illness

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 537 (Actual)
Dates: Start 2009-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Progression to diabetes | 6 monthly intervals for 2 years
  Prevention of type 2 diabetes in high-risk subjects by lifestyle modification

SECONDARY OUTCOMES:
Improvement in metabolic risk factors for diabetes and cardiovascular diseases and improvement in quality of life | two years
Acceptability of text messaging as tool to prevent diabetes. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Ambady Ramachandran, M.D, D.Sc, Principal Investigator — President, India Diabetes Research Foundation and Chairman & Managing Director, Dr.A.Ramachandran's Diabetes Hospitals; Desmond Geoffrey Johnston, MB Ch B, Ph.D, Principal Investigator — Professor of Clinical Endocrinology, Imperial College, London
Locations (1):
- Dr.Ambady Ramachandran, Chennai, Tamil Nadu, India

REFERENCES:
- [Background] Ramachandran A, Snehalatha C, Mary S, Mukesh B, Bhaskar AD, Vijay V; Indian Diabetes Prevention Programme (IDPP). The Indian Diabetes Prevention Programme shows that lifestyle modification and metformin prevent type 2 diabetes in Asian Indian subjects with impaired glucose tolerance (IDPP-1). Diabetologia. 2006 Feb;49:289-97. PMID: 16391903 Snehalatha C, Mary S, Joshi VV, Ramachandran A. Beneficial effects of strategies for primary prevention of diabetes on cardiovascular risk factors: results of the Indian Diabetes Prevention Programme. Diab Vasc Dis Res. 2008 Mar;5:25-9. PMID: 18398809 Murugesan N, Snehalatha C, Shobhana R, Roglic G, Ramachandran A. Awareness about diabetes and its complications in the general and diabetic population in a city in southern India. Diabetes Res Clin Pract. 2007 Sep;77:433-7. PMID: 17291622 Ramachandran A, Mary S, Yamuna A, Murugesan N, Snehalatha C. High prevalence of diabetes and cardiovascular risk factors associated with urbanization in India. Diabetes Care. 2008 May;31:893-8. PMID: 18310309 Ramachandran A. Epidemiology of diabetes in India--three decades of research. J Assoc Physicians India. 2005 Jan;53:34-8. Review. PMID: 15857011
- [Derived] Nanditha A, Jagannathan R, Sundaram S, Susairaj P, Shetty AS, Snehalatha C, Ian GF, Johnston DG, Ramachandran A. Combining Fasting Plasma Glucose with Gamma-glutamyl Transferase Improves the Sensitivity to Predict Incident Diabetes in Asian Indian Men with Impaired Glucose Tolerance. J Assoc Physicians India. 2014 Nov;62(11):18-22. PMID 26281475
- [Derived] Ram J, Selvam S, Snehalatha C, Nanditha A, Simon M, Shetty AS, Godsland IF, Johnston DG, Ramachandran A. Improvement in diet habits, independent of physical activity helps to reduce incident diabetes among prediabetic Asian Indian men. Diabetes Res Clin Pract. 2014 Dec;106(3):491-5. doi: 10.1016/j.diabres.2014.09.043. Epub 2014 Oct 25. PMID 25458326
- [Derived] Nanditha A, Ram J, Snehalatha C, Selvam S, Priscilla S, Shetty AS, Arun R, Godsland IF, Johnston DG, Ramachandran A. Early improvement predicts reduced risk of incident diabetes and improved cardiovascular risk in prediabetic Asian Indian men participating in a 2-year lifestyle intervention program. Diabetes Care. 2014 Nov;37(11):3009-15. doi: 10.2337/dc14-0407. Epub 2014 Sep 11. PMID 25216506
- [Derived] Hughes RC, Moore MP, Gullam JE, Mohamed K, Rowan J. An early pregnancy HbA1c >/=5.9% (41 mmol/mol) is optimal for detecting diabetes and identifies women at increased risk of adverse pregnancy outcomes. Diabetes Care. 2014 Nov;37(11):2953-9. doi: 10.2337/dc14-1312. Epub 2014 Sep 4. PMID 25190675
- [Derived] Ramachandran A, Snehalatha C, Ram J, Selvam S, Simon M, Nanditha A, Shetty AS, Godsland IF, Chaturvedi N, Majeed A, Oliver N, Toumazou C, Alberti KG, Johnston DG. Effectiveness of mobile phone messaging in prevention of type 2 diabetes by lifestyle modification in men in India: a prospective, parallel-group, randomised controlled trial. Lancet Diabetes Endocrinol. 2013 Nov;1(3):191-8. doi: 10.1016/S2213-8587(13)70067-6. Epub 2013 Sep 11. PMID 24622367